CLINICAL TRIAL: NCT07241143
Title: Comparison of the Efficacy and Safety of Extra-Peritoneal Tunneling Drain Fixation Versus Conventional Drain Insertion Following Anterior or Low Anterior Resection (ExPeTuD Trial): A Multi-Center Randomized Controlled Trial
Brief Title: Extra-Peritoneal Tunneling Versus Conventional Drain Fixation After Anterior or Low Anterior Resection
Acronym: ExPeTuD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yeungnam University Hospital (Other)
Collaborators: Konyang University Hospital (Other); Daegu Catholic University Medical Center (Other); Seoul National University Bundang Hospital (Other); Samsung Medical Center (Other); Seoul National University Hospital (Other); Severance Hospital (Other); Chungnam National University Hospital (Other); Chungbuk National University Hospital (Other); Keimyung University Dongsan Medical Center (Other); Pusan National University Yangsan Hospital (Other); Chonbuk National University Hospital (Other); Kyungpook National University Chilgok Hospital (Other); Yonsei University Yongin Severance Hospital (Unknown); Chonnam National University Hospital (Other); Ewha Womans University Seoul Hospital (Other); Soonchunhyang University Hospital (Other); Hallym University Dongtan Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Sung il Kang, Associate Professor, Yeungnam University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-08-031
Record Dates: First submitted 2025-11-13; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Rectal Diseases, Sigmoid Colon Disease; Rectal Cancer, Sigmoid Colon Cancer
Keywords: drain, anterior resection, low anterior resection
MeSH Terms: conditions — Rectal Diseases; Sigmoid Diseases; Rectal Neoplasms; Sigmoid Neoplasms

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group, randomized controlled design to compare two surgical techniques for pelvic drain insertion following anterior or low anterior resection for rectal cancer. Participants will be randomly assigned in a 1:1 ratio to either the extra-peritoneal tunneling (EPT) drain fixation group or the conventional drain insertion group. Randomization will be stratified by sex, preoperative chemoradiation status, and the anastomotic level relative to the peritoneal reflection to ensure balanced distribution of clinical factors.
Masking Description: All enrolled patients will undergo the same standard surgical and postoperative management, except for the method of drain placement. No masking will be applied because the surgical procedure is visibly different and performed intraoperatively. The trial will follow participants through postoperative recovery until drain removal and hospital discharge, with standardized imaging to assess drain position and detect anastomotic leakage. This design allows for direct comparison of efficacy and safety outcomes between the two techniques in real-world surgical settings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional drain insertion (Active Comparator): Participants undergo standard transperitoneal pelvic drain placement following anterior or low anterior resection.
  Interventions: Procedure: Conventional drain insertion
- EPT drain fixation (Experimental): Participants undergo pelvic drain placement using the extra-peritoneal tunneling (EPT) method following anterior or low anterior resection.
  Interventions: Procedure: EPT drain fixation

INTERVENTIONS:
Procedure: EPT drain fixation — Participants in this arm will receive pelvic drain placement using the extra-peritoneal tunneling (EPT) drain fixation method after anterior or low anterior resection for rectal cancer. The drain is then passed through this tunnel and positioned close to the anastomosis to maintain stable drainage and prevent displacement
  Arms: EPT drain fixation
Procedure: Conventional drain insertion — Participants in this arm will receive pelvic drain placement using the conventional transperitoneal method after anterior or low anterior resection for rectal cancer. In this standard technique, the drain is inserted directly through a lower abdominal port site (usually the left lower quadrant) into the pelvic cavity without creating an extraperitoneal tunnel
  Arms: Conventional drain insertion

SUMMARY:
The goal of this clinical trial is to learn whether the extra-peritoneal tunneling (EPT) drain fixation method works better and more safely than the conventional drain insertion method after rectal cancer surgery.

It will also learn about the safety and possible complications of the EPT technique.

The main questions it aims to answer are:

Does the EPT drain fixation method increase the success rate of conservative management (drain maintenance and/or antibiotics) when an anastomotic leak occurs?

Does the EPT method reduce the rate of drain displacement compared with the conventional method?

Are there any safety concerns or complications associated with the EPT method?

Researchers will compare EPT drain fixation to the conventional drain method to see which approach provides better outcomes after anterior or low anterior resection for rectal cancer.

Participants will:

Undergo anterior or low anterior resection for rectal cancer as part of their standard surgical treatment.

Be randomly assigned to either the EPT drain fixation group or the conventional drain group.

Receive the same postoperative care as usual, including follow-up imaging to monitor drain position and recovery.

Be observed for postoperative outcomes such as anastomotic leakage, drain position, and related complications until recovery.

This study will help determine whether securing the drain through an extra-peritoneal tunnel can prevent drain movement, improve early management of leakage, and enhance patient recovery after rectal surgery.

DETAILED DESCRIPTION:
resection for rectal cancer. Although prophylactic pelvic drainage has been widely used to detect early leakage and to prevent pelvic sepsis, recent randomized trials and meta-analyses have reported that routine drain placement provides no significant benefit in reducing postoperative morbidity. One possible reason is drain displacement, which occurs in up to 30-40% of cases, resulting in the drain being positioned far from the anastomotic site and losing its intended function.

The extra-peritoneal tunneling (EPT) drain fixation method is a new surgical technique designed to prevent drain displacement by creating an extraperitoneal tunnel that anchors the drain securely near the anastomosis. This technique is performed using the Drain-TG™ (DTG) device developed by JSR Medical (Daegu, Korea). Preliminary retrospective data have shown that the EPT technique dramatically reduces drain displacement (2.8% vs. 40% with conventional insertion, p < 0.001) and that, in patients who developed AL, the success rate of conservative management (drain maintenance and antibiotics only) exceeded 80%, compared with 43% in the conventional group.

The ExPeTuD trial is a prospective, multi-center, randomized controlled trial that aims to establish strong evidence for the efficacy and safety of the EPT drain fixation method. Patients undergoing anterior or low anterior resection with a predicted anastomosis ≤ 10 cm from the anal verge will be enrolled from approximately 20 tertiary hospitals across Korea. Participants will be randomized 1:1 to either the EPT group or the conventional drain group, stratified by sex, tumor level (above vs. below the peritoneal reflection), and preoperative chemoradiation status.

The primary outcome is the success rate of conservative management (drain maintenance and/or antibiotics) for AL according to drain insertion method. Secondary outcomes include:

Rate and timing of drain displacement (defined as > 3 cm separation from the anastomotic site on X-ray),

Drain-related complications (infection, pain, bleeding, or organ injury),

Time to diagnosis of AL and time to re-intervention,

Postoperative recovery outcomes such as ileus, hospital stay, and overall morbidity (Clavien-Dindo classification).

Radiologic monitoring (abdominal X-rays on postoperative days 2, 4, and 6) will be performed to assess drain position, and additional imaging will be conducted if AL is suspected. Standard postoperative care, including enhanced recovery after surgery (ERAS) protocols, will be applied equally to both groups.

A total of 596 participants (298 per arm) will be recruited, which accounts for an expected 6% AL rate after low anterior resection and ensures sufficient power for superiority testing. Interim analysis will be conducted once ≥ 9 AL events occur in each group to assess safety and trial feasibility.

If the EPT drain fixation method proves effective in maintaining drain position and improving conservative management success rates, it could reduce the need for reoperation, shorten hospital stay, and improve patient outcomes after rectal cancer surgery. This trial aims to provide robust clinical evidence supporting the adoption of the EPT technique as a standard method for pelvic drainage following proctectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo rectal resection (anterior resection or low anterior resection) with planned intraoperative drain placement.
* Expected anastomotic level ≤10 cm from the anal verge based on preoperative imaging or endoscopic evaluation.

Exclusion Criteria:

* Patients scheduled to undergo additional colonic resection (e.g., right hemicolectomy, transverse colectomy).
* Patients in whom no intraoperative drain placement is planned.
* Patients scheduled for permanent or end stoma formation (e.g., abdominoperineal resection or Hartmann's procedure).
* Patients with prior pelvic surgery (e.g., hysterectomy, prostatectomy, pelvic lymph node dissection) that may cause pelvic adhesions or anatomic distortion.
* Patients with ASA physical status IV or severe systemic disease expected to require postoperative intensive care unit (ICU) admission.
* Patients who decline to provide informed consent for study participation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Rate of successful conservative management in patients who developed an anastomotic leak | Within 60 days after diagnosis of anastomotic leak
  The success of conservative management is defined as resolution of the anastomotic leak without the need for reoperation or diversion. Success rates will be compared between patients managed with the Extra-Peritoneal Tunneling (EPT) drain fixation method and those with the conventional intraperitoneal drain placement.

SECONDARY OUTCOMES:
Incidence of drain displacement according to drain fixation method | Up to drain removal, an average of 7 days
  Drain displacement is defined as any unintended displacement of the drain from the originally intended position, confirmed by radiologic verification (X-ray or CT). Drain displacement is defined as a drain-to-anastomosis shortest distance exceeding 3 cm on an radiologic imaging compared with the immediate postoperative position. Incidence (%) of displacement will be compared between the Extra-Peritoneal Tunneling (EPT) and conventional drain fixation groups.
Time to drain displacement (days) | Up to drain removal, an average of 7 days
  Defined as the number of days from surgery to the date when drain displacement (drain-to-anastomosis shortest distance >3 cm on erect abdominal view) is first observed.
Incidence and types of drain-related complications according to drain fixation method | Up to drain removal, an average of 7 days
  Includes any adverse events directly related to the drain, such as infection at the insertion site, pain, skin irritation, etc.
Early detection of anastomotic leak (days from surgery to diagnosis) | Time to anastomotic leak, assessed up to 90 days after surgery
  Evaluates whether the use of EPT drain fixation facilitates earlier identification of anastomotic leak. Measured as the number of days from surgery to the confirmed diagnosis of anastomotic leak.
Interval between anastomotic leak diagnosis and reoperation (hours) | Time from leak diagnosis to reoperation, assessed up to 30 days after leak diagnosis
  Measures the time interval between the diagnosis of anastomotic leak and reoperation, including documentation of whether the reoperation occurred as an emergency or elective procedure.

CONTACTS AND LOCATIONS:
Overall Officials: SUNG IL KANG, M.D., Ph.D., Principal Investigator — Yeungnam University Hospital
Locations (1):
- Sung Il Kang, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
We have not yet determined whether individual participant data (IPD) will be shared. If sharing is approved, only de-identified IPD related to primary and key secondary outcomes will be made available.